CLINICAL TRIAL: NCT02388854
Title: Influence of WNT4 VEZT FSHB and SIRT1 Genetic Polymorphisms in the Pathogenesis of Endometriosis: a Case Control Study of the Sardinian Population
Brief Title: Influence of WNT4 VEZT FSHB and SIRT1 SNPs in Endometriosis: a Case Control Study of the Sardinian Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Influence of WNT4 VEZT FSHB and SIRT1 genetic polymorphiisms in the pathogenesis of endometriosis: a case control study of the Sardinian population, University of Cagliari
Other Study IDs: ENDOSNPs
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Polymorphism (Genetics); Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Endometriosis: Sardinian Women with diagnosis of endometriosis
  Interventions: Genetic: SNPs analysis with Sanger sequencing
- Controls: Healthy blood Sardinian donors
  Interventions: Genetic: SNPs analysis with Sanger sequencing

INTERVENTIONS:
Genetic: SNPs analysis with Sanger sequencing — Research of frequency of SNPs (WNT4, VEZT, FSHB and SIRT1 genes) in Sardinian women affected by endometriosis and controls

SUMMARY:
Endometriosis, defined as the presence of endometrial tissue outside the uterine cavity, affects 6-10% of the general population of women in childbearing age.

The pathogenesis of the disease is unknown. The purpose of this study is to evaluate the influence of certain polymorphisms of genes WNT4, VEZT, FSHB, known to be involved in molecular mechanisms associated with phenomena of proliferation and development of endometriotic lesions, and SIRT1, that based on metabolomics studies, could hypothetically have a role in the pathogenesis of the disease. The study focus on the Sardinian population, known to have unique genetic characteristics due to geographical isolation.

DETAILED DESCRIPTION:
Endometriosis is a benign estrogen-dependent disease characterized by the presence of endometrial tissue in its glandular and stromal components in locations other than the uterine cavity . Represents one of the most common gynecological, chronic inflammatory diseases of women of reproductive age, affecting approximately 10% of the female population, although this estimate may be lower than the real data considering the heterogeneity of the clinical manifestations of the disease and the tendency to therefore be underdiagnosed . Endometriosis is often associated with infertility and severe pain symptomatology including chronic pelvic pain, dyspareunia and dysmenorrhea. Despite numerous studies, the pathogenesis of the disease is still unknown. Studies on family aggregation and twins have given prominence to the genetic component, demonstrating how the genetic structure inherited from an individual influences 51% of the predisposition to develop endometriosis in life. A great deal of work has involved the identification of different gene polymorphisms able to help explain the susceptibility to the development of endometriosis, often with conflicting results . Genome-wide association studies (GWAS) and related meta-analyzes have led to the identification of disease risk loci by providing new insights into potential molecular pathways involved in endometriosis. At present, 19 independent single-nucleotide polymorphisms (SNPs) have been validly associated with endometriosis, explaining 5.19% of the variance of the disease.In particular, a recent study investigated three of these SNPs on the Greek population: rs7521902, rs10859871 and rs11031006, mapped respectively on the WNT4, VEZT and FSHB genes, highlighting a significant association with endometriosis. The WNT4 gene, located on chromosome 1, codes for a fundamental protein in the development of the female reproductive system . The expression of WNT4 has also been demonstrated at the level of the normal peritoneum suggesting a possible metaplastic hypothesis in promoting the transformation of peritoneal cells into endometriotic cells using pathways involved in the development of female genital tracts. Moreover WNT4 is equally expressed in the eutopic endometrium during the proliferative and secretory phases; variants of this gene could hypothetically contribute to abnormal growth of endometrial cells in ectopic sites. VEZT is a gene located on chromosome 12 and coding for vezatin, an important component of the cadherin-catenin complex which is essential for the formation and maintenance of adherent joints. The protein is expressed in most epithelial cells and is crucial for the formation of cell-cell contact junctions. The expression of VEZT is altered in the endometrium of patients with endometriosis and is an excellent candidate for having a causal role in endometriosis. In particular, the rs10859871 polymorphism was associated with an increase in the expression of this gene.The FSHB gene, located on chromosome 11, codes for the hormone-specific subunit b of the stimulating follicle hormone (FSH), a key promoter of ovarian follicle growth and estrogen production. The extended GWAS of the Sapkota group identifies a significant association between the rs11031006 polymorphism and the risk of endometriosis.

The metabolomic profile in patients affected by endometriosis have identified beta-hydroxybutyrate (bOHB) as a significantly increased metabolite in affected patients. The bOHB is a ketonic body that acts as an energy carrier from adipocytes to peripheral tissues. However, it plays a heterogeneous role in cellular signaling and regulation of gene expression. Several enzymes involved in the generation of ketone bodies from lipids are both acetylated and succinylated and target a group of enzymatic activity proteins that act as NAD-dependent deacylases: sirtuins. Sirtuins have recently been studied for their involvement in the field of female reproductive function. Among these, sirtuine 1, SIRT1, acts as histone-deacetylase and is implicated in innumerable phenomena such as the regulation of gene transcription, aging, stress resistance, apoptosis, energy efficiency. Furthermore, SIRT1 plays an important role in regulating the expression of inflammatory cytokines in endometriotic stromal cells. The SIRT1 gene, located on chromosome 10, is over-expressed in the eutopic endometrium of women with endometriosis and is probably involved in the pathogenesis of endometriosis. SIRT1 controls among other things the acetylation of a fork transcription factor involved in the pathway metabolic synthesis of ketone bodies, FOXA2, in turn involved in the phenomena of proliferation and migration of endometriotic cells. Some SSPs of the SIRT1 gene are associated with insults from oxidative stress capable of inducing an abnormal proliferation of endometrial cells (k endometrium).

The study aims to verify the possible association between the presence of certain polymorphisms of genes known to have a hypothetical role in the pathogenesis of endometriosis and the development of this disease in the population of Sardinian origin.

The study will be carried out by molecular typing of the following single substitution polymorphisms (SNPs): rs7521902, rs10859871, rs11031006, rs2273773, mapped respectively in the WNT4, VEZT, FSHB and SIRT1 genes.

In this work will be described the frequency of alleles, genotypes and haplotypes of these SNPs among Sardinian women and will be evaluated their impact on susceptibility to the development of endometriosis.

The molecular-biological analyzes of single-substitution polymorphisms will be carried out starting from whole blood, taken, subject to informed consent, to exclusively Sardinian patients.

The investigators have chosen to limit the study only to patients originating from Sardinia, taking advantage of the peculiarity of this land, which can be considered a genetic macro-isolate. The genetic analysis of complex traits is in fact simplified in isolated populations like the Sardinian one, in which inbreeding and "founding effect" reduce the genetic diversity of complex and polygenic diseases such as endometriosis which can, in this way, be studied more easily.The goal is to identify a genetic characterization that can be used for the non-invasive diagnosis of the disease

ELIGIBILITY:
Inclusion Criteria (cases):

* endometriosis diagnosis (clinic, ultrasound or histological)
* women of Sardinian origin

Inclusion Criteria (controls):

* no signs of endometriosis
* women of Sardinian origin

Exclusion Criteria (cases and controls):

* women of non-Sardinian origin
* patients unable to provide written informed consent or to follow the procedures provided by the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sardinian women with or without diagnosis of endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of Single Nucleotide Polymorphisms of WNT4, VEZT, FSHB and SIRT1 in Sardinian women with and without endometriosis diagnosis | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cagliari,Obstetrics and Gynecological Department,, Monserrato, Cagliari, Italy

REFERENCES:
- [Background] Matalliotakis M, Zervou MI, Matalliotaki C, Rahmioglu N, Koumantakis G, Kalogiannidis I, Prapas I, Zondervan K, Spandidos DA, Matalliotakis I, Goulielmos GN. The role of gene polymorphisms in endometriosis. Mol Med Rep. 2017 Nov;16(5):5881-5886. doi: 10.3892/mmr.2017.7398. Epub 2017 Aug 29. PMID 28901453
- [Background] Sapkota Y, Steinthorsdottir V, Morris AP, Fassbender A, Rahmioglu N, De Vivo I, Buring JE, Zhang F, Edwards TL, Jones S, O D, Peterse D, Rexrode KM, Ridker PM, Schork AJ, MacGregor S, Martin NG, Becker CM, Adachi S, Yoshihara K, Enomoto T, Takahashi A, Kamatani Y, Matsuda K, Kubo M, Thorleifsson G, Geirsson RT, Thorsteinsdottir U, Wallace LM; iPSYCH-SSI-Broad Group; Yang J, Velez Edwards DR, Nyegaard M, Low SK, Zondervan KT, Missmer SA, D'Hooghe T, Montgomery GW, Chasman DI, Stefansson K, Tung JY, Nyholt DR. Meta-analysis identifies five novel loci associated with endometriosis highlighting key genes involved in hormone metabolism. Nat Commun. 2017 May 24;8:15539. doi: 10.1038/ncomms15539. PMID 28537267